CLINICAL TRIAL: NCT01521559
Title: A Double-Masked, Randomized, Active-Controlled Study of the Efficacy, Safety, and Tolerability of Intravitreal Administration of VEGF Trap-Eye (Intravitreal Aflibercept Injection [IAI]) in Patients With Macular Edema Secondary to Branch Retinal Vein Occlusion
Brief Title: Study to Assess the Clinical Efficacy and Safety of Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) in Patients With Branch Retinal Vein Occlusion (BRVO)
Acronym: VIBRANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGFTe-RVO-1027
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Macular Laser Photocoagulation Treatment (Control) (Sham Comparator): Participants will receive macular laser treatment at Baseline and then according to laser re-treatment criteria up to week 24. Participants will receive treatment with Intravitreal Aflibercept Injection (IAI) starting at week 24 if they met rescue criteria. Treatment with IAI once initiated was 3 initial monthly doses followed by Q8 week dosing.
  Interventions: Procedure: Macular Laser Photocoagulation
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4 (Experimental): Participants will receive 2 milligrams (mg) Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) through week 24 followed by injections every 8 weeks (2Q8) through week 48. Participants in this group may receive laser rescue at week 36.
  Interventions: Drug: Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)

INTERVENTIONS:
Procedure: Macular Laser Photocoagulation
  Arms: Macular Laser Photocoagulation Treatment (Control)
Drug: Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
  Arms: Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) 2Q4

SUMMARY:
This is a phase III, double-masked, randomized, active-controlled, parallel-group, 52-week study to assess the efficacy and safety of Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) compared to laser treatment in patients with macular edema secondary to BRVO.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria include, but are not limited to:

1. Adults ≥ 18 years of age with foveal center-involved macular edema (ME) secondary to BRVO diagnosed within 12 months before the screening visit
2. ETDRS BCVA: letter score of 73 to 24 (20/40 to 20/320) in the study eye at screening and at day 1
3. Provide signed informed consent

Exclusion Criteria:

The following exclusion criteria include, but are not limited to:

1. Current bilateral manifestation of BRVO
2. Uncontrolled glaucoma defined as ≥ 25 mmHg on optimal medical regimen, or previous filtration surgery in either the study eye or the fellow eye
3. Insufficient clearing of macular hemorrhage that would prevent the patient from receiving laser treatment safely on day 1 (patients that meet this criterion may be rescreened once the macular hemorrhage resolves)
4. Uncontrolled diabetes mellitus (DM)
5. Previous use of intraocular corticosteroids or anti-angiogenic drugs in the study eye
6. Use of periocular corticosteroids in the study eye within 3 months before day 1
7. Use of intraocular or periocular corticosteroids or anti-angiogenic drugs in the fellow eye within 3 months before day 1
8. Previous administration of systemic anti-angiogenic medications
9. Panretinal scatter photocoagulation, sector laser photocoagulation, or macular grid photocoagulation in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (56):
- United States (45):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - La Jolla, California
  - Mountain View, California
  - Palm Desert, California
  - Sacramento, California
  - Colorado Springs, Colorado
  - Fort Myers, Florida
  - Miami, Florida
  - Plantation, Florida
  - Stuart, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Baltimore (2 Locations), Maryland
  - Hagerstown, Maryland
  - Boston (2 Locations), Massachusetts
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Southfield, Michigan
  - Florissant, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Teaneck, New Jersey
  - Orchard Park, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Kingston, Pennsylvania
  - West Mifflin, Pennsylvania
  - Florence, South Carolina
  - Ladson, South Carolina
  - West Columbia, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Fort Worth, Texas
  - Harlingen, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Canada (4):
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Mississauga, Ontario
  - Toronto, Ontario
- Japan (7):
  - Urayasu-shi, Chiba
  - Fukushima, Fukushima
  - Amagasaki, Hyōgo
  - Kagoshima, Kagoshima-ken
  - Kyoto, Kyoto
  - Osaka, Osaka
  - Hamamatsu, Shizuoka

REFERENCES:
- [Derived] Shalchi Z, Mahroo O, Bunce C, Mitry D. Anti-vascular endothelial growth factor for macular oedema secondary to branch retinal vein occlusion. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD009510. doi: 10.1002/14651858.CD009510.pub3. PMID 32633861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with macular edema secondary to branch retinal vein occlusion (BRVO) involving the center of the macula in the study eye were eligible to participate in the study.
Pre-assignment Details: Of 281 participants who were screened for inclusion in the study, 183 were enrolled (started) and 183 received treatment.
Groups:
- Macular Laser Photocoagulation Treatment (Control): Participants received macular laser treatment at Baseline and then according to laser re-treatment criteria up to week 24. Participants received treatment with Intravitreal Aflibercept Injection (IAI) starting at week 24 if they met rescue criteria. Treatment with IAI once initiated was 3 initial monthly doses followed by Q8 week dosing.
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321): Participants received 2 milligrams (mg) Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) through week 24 followed by injections every 8 weeks (2Q8) through week 48. Participants in this group could receive laser rescue at week 36.
Period: Overall Study
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Started | 92 | 91
Completed Week 24 | 83 | 85
Completed Week 52 | 77 | 73
Completed | 77 | 73
Not Completed | 15 | 18
Not completed — Adverse Event | 0 | 4
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 9 | 11
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Other | 1 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All enrolled subjects who received any investigational product, had a baseline best corrected visual acuity (BCVA) assessment, and at least 1 post-baseline BCVA assessment.
Groups:
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321): Participants received 2 mg Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) through week 24 followed by injections every 8 weeks (2Q8) through week 48. Participants in this group could receive laser rescue at week 36.
- Total: Total of all reporting groups
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) | Total
Number analyzed (Participants) | 90 | 91 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.37) | 67.0 (10.41) | 65.5 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 47 | 83
  Male | 54 | 44 | 98

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Gained at Least 15 Letters in Best Corrected Visual Acuity (BCVA) at Week 24 - LOCF
Description: Best corrected visual acuity (BCVA) was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at every visit from baseline through week 24. Last observation carried forward (LOCF) method was used to impute missing data.
Time Frame: Baseline to week 24
Population: FAS
Measure: Number; unit: participants
Groups:
- Macular Laser Photocoagulation Treatment (Control): Participants received macular laser treatment at Baseline and then according to laser re-treatment criteria up to week 24.
- Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321): Participants received 2 mg Intravitreal Aflibercept Injection (IAI) every 4 weeks (2Q4) through week 24.
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Number analyzed (Participants) | 90 | 91
participants | 24 | 48
Statistical Analysis 1: Comparison: Macular Laser Photocoagulation Treatment (Control) vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321); Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel — P-value was calculated using 2-sided Cochran-Mantel-Haenszel test adjusted by regions (Japan vs North America) and baseline Best Corrected Visual Acuity (BCVA ≤20/200 and BCVA >20/200); Mean Difference (Net) = 26.6, 95% CI 2-sided [13.0 to 40.1] — Difference was IAI group minus laser group; Difference and confidence interval were calculated using Mantel-Haenszel weighting scheme adjusted by regions (Japan vs North America) and baseline BCVA (BCVA ≤20/200 and BCVA >20/200)

2. Secondary Outcome: Change From Baseline to Week 24 in BCVA Score - LOCF
Description: Best corrected visual acuity (BCVA) was assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol at every visit from baseline through week 24 - Last observation carried forward (LOCF) method was used to impute missing data.
Time Frame: Baseline to Week 24
Population: FAS
Measure: Mean (Standard Deviation); unit: letters correctly read
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Number analyzed (Participants) | 90 | 91
letters correctly read | 6.9 (12.91) | 17.0 (11.88)
Statistical Analysis 1: Comparison: Macular Laser Photocoagulation Treatment (Control) vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321); Difference was IAI group minus laser group. P-value, Point estimate and 95% confidence interval (CI) were based on an analysis of covariance (ANCOVA) model with baseline measurement as covariate and treatment group, region, and baseline Best Corrected Visual Acuity (BCVA ≤20/200 and BCVA >20/200) as fixed factors; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = 10.5, 95% CI 2-sided [7.1 to 14.0]

3. Secondary Outcome: Change From Baseline in Central Retinal Thickness (CRT) at Week 24 - LOCF
Description: CRT was evaluated at every visit from baseline through week 24 using spectral domain Optical Coherence Tomography (OCT).
Time Frame: Baseline to week 24
Population: FAS
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Number analyzed (Participants) | 90 | 91
microns | -128.0 (195.02) | -280.5 (189.7)
Statistical Analysis 1: Comparison: Macular Laser Photocoagulation Treatment (Control) vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321); Difference was IAI group minus laser group; P-value, Point estimate, and 95% CI, were based on an ANCOVA model with baseline measurement as covariate and treatment group, region, and baseline Best Corrected Visual Acuity (BCVA ≤20/200 and BCVA >20/200) as fixed factors; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Net) = -148.6, 95% CI 2-sided [-179.8 to -117.4]

4. Secondary Outcome: Change From Baseline in the National Eye Institute Visual Function Questionnaire - 25 (NEI VFQ-25) Questionnaire Total Score at Week 24 - LOCF
Description: The NEI VFQ-25 total score ranges from 0-100 with a score of 0 being the worst outcome and 100 being the best outcome. The NEI VFQ questionnaire is organized as a collection of subscales that are all scored from 0-100. Near activities are defined as reading ordinary print in newspapers, performing work or hobbies requiring near vision, or finding something on a crowded shelf.
Time Frame: Baseline to week 24
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Number analyzed (Participants) | 87 | 88
scores on a scale | 6.3 (12.34) | 7.7 (11.08)
Statistical Analysis 1: Comparison: Macular Laser Photocoagulation Treatment (Control) vs Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321); [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0833, ANCOVA; Mean Difference (Net) = 2.6, 95% CI 2-sided [-0.3 to 5.5]

ADVERSE EVENTS:
Time Frame: Through Week 52 (end of study)
Description: The safety analysis set (SAF) included all enrolled participants who received any investigational product; it is based on the treatment received (as treated).
Arm/Group | Macular Laser Photocoagulation Treatment (Control) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321)
Serious Adverse Events (participants affected / at risk) | 10/92 | 13/91
Other Adverse Events (participants affected / at risk) | 30/92 | 25/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macular Laser Photocoagulation Treatment (Control) (N=92) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) (N=91)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cataract traumatic (Injury, poisoning and procedural complications) | 0 | 1 — Study eye
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Delayed haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hernia (General disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 2
Presyncope (Nervous system disorders) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transaminases increased (Investigations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macular Laser Photocoagulation Treatment (Control) (N=92) | Intravitreal Aflibercept Injection (IAI;EYLEA®;BAY86-5321) (N=91)
Blood pressure increased (Investigations) | 5 | 4
Bronchitis (Infections and infestations) | 2 | 6
Conjunctival haemorrhage (Eye disorders) | 14 | 22 — Study eye
Eye irritation (Eye disorders) | 1 | 7 — Study eye
Eye pain (Eye disorders) | 7 | 5 — Study eye
Hypertension (Vascular disorders) | 15 | 9
Nasopharyngitis (Infections and infestations) | 8 | 8
Urinary tract infection (Infections and infestations) | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Without the prior written agreement of the Sponsor, the Institution (I) shall not publish, submit or present for publication, directly or indirectly, any Manuscript (M) prior to publication of an article in a peer-reviewed scientific journal summarizing data generated by all Study centers, unless no such article is so published before the first anniversary of the finalization of the clinical study report, in which case the (I) may publish or submit for publication a (M) without further delay.